CLINICAL TRIAL: NCT03142295
Title: Safety and Tolerability of Controlled Human Urine Transfusion for Urinary Tract Infection Prevention (SHUTUP): a Pilot Study
Brief Title: Controlled Human Urine Transfusion for UTI
Acronym: SHUTUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, ImroVlasveld, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL60330.058.16
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Recurrent Urinary Tract Infection; Safety Issues
Keywords: Urine transfusion; Recurrent urinary tract infection; Urinary microbiota
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: prospective, open label pilot clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urine transfusion (Experimental): Intervention: Two transfusions of 100 ml of urine within 5 days by transurethral catheterization after an antibiotic free interval of 3 days.
  Interventions: Procedure: urine transfusion

INTERVENTIONS:
Procedure: urine transfusion — Two transfusions of 100 ml of urine within 5 days by transurethral catheterization after an antibiotic free interval of 3 days.

SUMMARY:
The primary objective of this pilot study is to investigate the safety and tolerability of controlled human urine transfusion in female patients with recurrent UTI's.

Seconday and exploratory objectives are to evaluate the diversity of the urine microbiome after urine transfusion, to assess the longevity of changes in the urine microbiome in patients after urine transfusion over a period of 6 months and to assess the frequency of UTI's after the transfusion.

DETAILED DESCRIPTION:
Recurrent urinary tract infections (UTIs) are the most common bacterial infections in nursing homes, in acute care and the general practice. Increasing antibiotic resistance of enterobacteriaciae poses a challenge to the treatment of UTIs. Unlike previously thought, the bladder is colonized with bacteria, which together form the urine microbiome. Recurrent urinary tract infections are associated with a decreased urinary microbiota diversity, potentially making recolonization by bacterial interference in the bladder an alternative therapy for UTI. Pioneering studies showed that local bacterial interference in the bladder can be performed safely and has potential as prophylactic intervention.

We now propose to expand this bacterial interference to a polymicrobial inoculum to increase adherence of the donor microbiome and as such expand the prophylactic effect. This pilot trial will investigate the safety and tolerability of urine transfusion from healthy donors to the bladders of patients with recurrent UTIs.

The primary objective of this pilot study is to investigate the safety and tolerability of controlled human urine transfusion in female patients with recurrent UTI's.

Secondary and exploratory objectives are to evaluate the diversity of the urine microbiome after urine transfusion, to assess the longevity of changes in the urine microbiome in patients after urine transfusion over a period of 6 months and to assess the frequency of UTI's after the transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Subject is premenopausal, aged ≥ 18 and ≤45 years
* Subject had recurrent UTI's (≥3 documented UTI's in the last year with documented symptom-free interval of at least 2 weeks) following the definition of a urinary tract infection: the presence of significance bacteruria (10^3 CFU/ml or more), pyuria and fever plus one or more of the following signs and symptoms: suprapubic or flank discomfort, dysuria, bladder spasms or pollakiuria
* Subject has a documented urinary tract infection (see definition), for which oral antibiotic therapy has been initiated.
* Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
* Subject is able to communicate well with the investigators and is available to attend all study visits.
* Subject has signed informed consent.
* Subject will remain available during the first 3 weeks of the study period (recruiting, intervention and first follow-up).

Exclusion Criteria:

* Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, immune-deficient, psychiatric and other disorders, which could compromise the health of the recipient during the study. These include, but are not limited to, any of the following: positive HIV, HBV or HCV screening tests; the use of immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.
* Documented vesico-urethral reflux
* Documented urinary retention > 100 milliliters post-void residual urine
* Anatomic urogenital abnormalities
* Urolithiasis
* Nephrostomy catheters
* Extra-urogenital infections that require prolonged antibiotic therapy
* Pregnancy
* Use of probiotics and or cranberry juice
* Allergy or intolerance for multiple common prescribed antibiotics
* Carriage of multi drug resistant organisms in faeces and/or urine without regular antibiotic treatment options

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-06-24 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety | 6 months
  The cumulative number of possibly, probably or definitely related adverse events within 6 months of controlled human urine transfusion

SECONDARY OUTCOMES:
Diversity of the urine microbiome after urine transfusion | 6 months
  Change in Shannon diversity index of the bladder microbiome before and after urine transfusion
The composition of the urine microbiome before and after urine transfusion | 6 months
  Percentage of the total microbiome occupied per genus by 16S sequencing
Frequency of UTIs after urine transfusions | 6 months
  The number of UTIs during the follow-up period of 6 months after the urine transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Imro Vlasveld, MD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No